CLINICAL TRIAL: NCT05608694
Title: MRI Screening in Men at High Risk of Developing Prostate Cancer
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Chicago (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Factorial | Masking: None | Purpose: Screening
Other Study IDs: IRB20-0038
Record Dates: First submitted 2022-10-10; First posted 2022-11-08 (Actual); Last update posted 2025-01-31 (Actual); Status verified 2025-01

CONDITIONS: Prostate Cancer Screening

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- High Risk- Positive Germline Mutation (n=40): (Other): Men who harbor known germline mutations that have been associated with an increased risk of prostate cancer and aggressive disease (e.g. BRCA2, ATM, PALB2, etc.) with or without a known family history of prostate cancer.
  Interventions: Other: Prostate MRI
- High Risk- High GRS (n=40): (Other): Men who harbor significantly increased disease risk based upon genetic risk score (GRS) value >1.5 with or without a known family history of prostate cancer.
  Interventions: Other: Prostate MRI
- High Risk- Family History (n=45): (Other): Men with a family history of prostate cancer in at least one sibling, father, uncle, or grandfather but no known increased genetic risk of prostate cancer (has no pathogenic or likely pathogenic mutation along with a low genetic risk score (GRS<1.5).
  Interventions: Other: Prostate MRI
- Low Risk (n=125): (Other): No known germline mutation, low genetic risk score (GRS <1.5), and no known family history of prostate cancer.
  Interventions: Other: Prostate MRI

INTERVENTIONS:
Other: Prostate MRI — Group placement is determined by GRS score, Family history, and germline testing

SUMMARY:
The purpose of this study is to determine whether or not Magnetic Resonance Images (MRI) will identify high-grade cancers earlier and more frequently in men at high risk of developing prostate cancer.

DETAILED DESCRIPTION:
In this study the study team hypothesizes MR images will identify high-grade cancers earlier and more frequently in men at high risk of developing prostate cancer. Subjects will receive gadolinium (intravenous contrast agent) as part of their research MRI exam. While the deposition of gadolinium (Gd) has been demonstrated in numerous studies, the clinical consequences of Gd deposition are unknown. Gd enhanced MRI scans provide crucial medical information regarding prostate and prostate cancer imaging and contrast-enhanced images are a component of all guidelines and the PIRADS scoring system. The study team will compare baseline prostate MR images of men at high risk of developing prostate cancer to those without an identifiable predisposition and evaluate the role of a GRS in screening men with at elevated risk of being diagnosed with prostate cancer.

ELIGIBILITY:
Inclusion Criteria:

* Male age 18 and older
* No known history of prostate cancer
* No previous prostate resection or ablation (e.g. TURP, photovaporization)

Exclusion Criteria:

* Unable to tolerate MRI due to metal fragments or claustrophobia
* Lack of a rectum
* Hip arthroplasty

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 250 (Estimated)
Dates: Start 2022-03-02 (Actual); Primary Completion 2037-03-01 (Estimated); Study Completion 2039-03-01 (Estimated)

PRIMARY OUTCOMES:
Proportion of patients with high grade prostate cancer detection. | Every 3 years up to 15 years
  MRI results will be collected every 3 years for 15 years until high grade prostate cancer is detected as defined as Gleason greater than or equal to 7 (Grade Group 2).

CONTACTS AND LOCATIONS:
Overall Officials: Scott Eggener, MD, Principal Investigator — University of Chicago
Locations (2):
- United States (2):
  - University of Chicago, Chicago, Illinois
  - NorthShore University Health System - Glenbrook Hospital, Glenview, Illinois

REFERENCES:
- [Background] Fazekas T, Shim SR, Basile G, Baboudjian M, Koi T, Przydacz M, Abufaraj M, Ploussard G, Kasivisvanathan V, Rivas JG, Gandaglia G, Szarvas T, Schoots IG, van den Bergh RCN, Leapman MS, Nyirady P, Shariat SF, Rajwa P. Magnetic Resonance Imaging in Prostate Cancer Screening: A Systematic Review and Meta-Analysis. JAMA Oncol. 2024 Jun 1;10(6):745-754. doi: 10.1001/jamaoncol.2024.0734. PMID 38576242
- [Background] Hugosson J, Godtman RA, Wallstrom J, Axcrona U, Bergh A, Egevad L, Geterud K, Khatami A, Socratous A, Spyratou V, Svensson L, Stranne J, Mansson M, Hellstrom M. Results after Four Years of Screening for Prostate Cancer with PSA and MRI. N Engl J Med. 2024 Sep 26;391(12):1083-1095. doi: 10.1056/NEJMoa2406050. PMID 39321360
- [Background] Bjornebo L, Discacciati A, Falagario U, Vigneswaran HT, Jaderling F, Gronberg H, Eklund M, Nordstrom T, Lantz A. Biomarker vs MRI-Enhanced Strategies for Prostate Cancer Screening: The STHLM3-MRI Randomized Clinical Trial. JAMA Netw Open. 2024 Apr 1;7(4):e247131. doi: 10.1001/jamanetworkopen.2024.7131. PMID 38648061